CLINICAL TRIAL: NCT02068612
Title: Enhancing Function in Later Life: Exercise and Functional Network Connectivity
Acronym: FORCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Angela Bryan, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01AG043452-01A1 (NIH)
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Aging
Keywords: Executive function,; cardiovascular fitness,; cognitive function

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MICT + IT (Experimental): Moderate Intensity Continuous Training+Interval Training
  Interventions: Behavioral: Moderate Intensity Continuous Training+Interval Training
- LICT (Active Comparator): Low Intensity Continuous Training
  Interventions: Behavioral: Low Intensity Continuous Training

INTERVENTIONS:
Behavioral: Moderate Intensity Continuous Training+Interval Training
  Other Names: MICT+IT
  Arms: MICT + IT
Behavioral: Low Intensity Continuous Training
  Other Names: LICT
  Arms: LICT

SUMMARY:
Physiological and neurocognitive changes experienced as a result of increasing age may influence socioemotional functioning and economic behaviors, yet, the mechanisms through which these changes occur are not well understood. Studies have also shown that aerobic exercise may protect against age-related cognitive decline in other domains. This research is designed to test the hypothesis that aerobic exercise will enhance social, emotional and economic functioning in older adults, and that these effects will occur via the effect of exercise on neurocognitive structure and function assessed via magnetic resonance imaging (MRI). Advancing our knowledge of the mechanisms that influence emotional, social and economic functioning could inform the development of targeted treatments and prevention programs for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-35 for younger adults, and age 60 or over for older adults
* Sedentary (i.e., < 60 minutes per week of moderate physical activity in the past 6-months)
* Able to make fewer than 3 errors on the Pfeiffer Mental Status192
* Willing to accept random assignment to condition (older adults)
* Physically capable of safely engaging in moderate exercise activity (i.e., no injuries, physical impairments, or pre-existing contraindications) as assessed by a study physician
* Able to successfully complete a maximal exercise test without evidence of cardiac or other abnormalities
* Planning to remain in the Boulder-Denver metro area for the next 4 months (older adults)

Exclusion Criteria:

* Are a heavy smoker (>20 pack years)
* Are diabetic
* Have a body size exceeding the capacity of the magnetic resonance imaging machine (approximately 23" in diameter)
* Are on antipsychotic medications
* Are currently under treatment for any psychiatric disorder, including clinical depression, Alzheimer's, or dementia
* Are currently pregnant
* Have magnetic resonance imaging contraindications (i.e., non-removable metallic implants, claustrophobia, traumatic brain injury, current pregnancy, etc.)

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2014-04; Primary Completion 2018-11-13 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Cognitive Function | 4 months
  1. Functional connectivity is measured via having participants lie in a magnetic resonance imaging scanner and passively stare at a centrally-positioned fixation crosshair for 8 min while their brain activity is recorded.
  2. Executive function will be measured with 3 tasks characterized by the three domains of executive function: updating, shifting, and inhibition. For updating, we will utilize the Keep Track task,for shifting, we will use the Category Switch Task, and for inhibition we will use the Stroop task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

REFERENCES:
- [Derived] Gust CJ, Martin-Willett R, Gibson LP, Giordano G, Seals DR, Bryan AD. Effects of aerobic exercise of different intensities on the social, emotional, and financial functioning of healthy older adults: results from a 16-week exercise randomized control trial. Geroscience. 2025 Apr 21. doi: 10.1007/s11357-025-01655-0. Online ahead of print. PMID 40259150
- [Derived] Martin-Willett R, Morris B, Wilcox R, Giordano G, Andrews-Hanna J, Banich M, Bryan AB. The influence of a 16-week exercise program, APOE status, and age on executive function task performance: A randomized trial. Exp Gerontol. 2021 Sep;152:111431. doi: 10.1016/j.exger.2021.111431. Epub 2021 May 29. PMID 34062261
- [Derived] Martin-Willett R, Ellingson JE, Fries J, Helmuth T, Karoly H, Giordano G, Calhoun VD, Bryan AD. Few Structural Brain Changes Associated With Moderate-Intensity Interval Training and Low-Intensity Continuous Training in a Randomized Trial of Fitness and Older Adults. J Aging Phys Act. 2021 Jun 1;29(3):505-515. doi: 10.1123/japa.2019-0352. Epub 2020 Dec 2. PMID 33271506
- [Derived] YorkWilliams SL, Gibson LP, Gust CJ, Giordano G, Hutchison KE, Bryan AD. Exercise Intervention Outcomes with Cannabis Users and Nonusers Aged 60 and Older. Am J Health Behav. 2020 Jul 1;44(4):420-431. doi: 10.5993/AJHB.44.4.5. PMID 32553024

DOCUMENTS (2):
  • Informed Consent Form: Older Adult Consent Form (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT02068612/ICF_000.pdf
  • Informed Consent Form: Young Adult Consent Form (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT02068612/ICF_001.pdf